CLINICAL TRIAL: NCT02045433
Title: A Phase II Study for Stereotactic Body Radiation Therapy (SABR) for Definitive Treatment of Locally Advanced Cervical Cancer (LACC)
Brief Title: Stereotactic Body Radiation Therapy (SABR) for Definitive Treatment of Locally Advanced Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely closed due to unacceptable toxicity.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 082013-064
Record Dates: First submitted 2014-01-14; First posted 2014-01-24 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2019-09

CONDITIONS: Locally Advanced Cervical Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SABR Boost Therapy (Experimental)
  Interventions: Radiation: SABR Boost Therapy

INTERVENTIONS:
Radiation: SABR Boost Therapy — 1. Initial Pelvic (+/- Para-aortic) fractionated external beam Radiation with 45 Gy to combined PTV with a boost to 55Gy for PET positive/CT enlarged nodes;
  2. Image Guided Hypofractionated Radiation Treatment boost to Cervix High risk CTV/PTV 28GY/4 fx.
  Patients will receive 4 fractions of 7 Gy each via stereotactic body radiation as boost therapy to a volume that encompasses the cervical tumor. A minimum of 40 hours should separate each treatment.

SUMMARY:
The purpose of this study is to determine whether SABR boost therapy is effective in women with locally advanced cervical cancer without increased risk of acute gastrointestinal (GI) or genitourinary (GU) toxicity.

DETAILED DESCRIPTION:
Patients enrolled in this study will receive 45 Gray (Gy) in 25 fractions of intensity modulated external beam radiation therapy + weekly cisplatinum . Following the completion of Intensity Modulated Radiation Therapy (IMRT), patients will receive 28 Gy in 4 fractions using stereotactic body radiation therapy techniques.

ELIGIBILITY:
Inclusion Criteria:

1 Locally Advanced stage Cervical Cancer 2. Zubrod performance status 0-2 3. Negative urine or serum pregnancy test for women of child-bearing potential 4. Agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment 5. Not a candidate for intracavitary brachytherapy

Exclusion Criteria:

1. Pregnancy
2. Concurrent untreated cancer excluding non-Melanoma skin cancer
3. Previous pelvic radiation
4. Active Inflammatory Bowel disease, Collagen vascular disease - systemic lupus erythematosus (SLE), scleroderma
5. Age <18
6. Unable to consent for study
7. Severely immunocompromised patients ( such as Transplant , on immunosuppressive drugs)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 16 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Albuquerque, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SABR Boost Therapy: SABR Boost Therapy for cervix cancer
Period: Overall Study
Arm/Group | SABR Boost Therapy
Started | 16
Completed | 15 (Study was Prematurely ended due to toxicity)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Image Guided Hypfractioned Radiation Treatment: Typically, only 1-5 fractions are used for Image Guided Hypofractionated RadiationTreatment depending on the tolerance of adjacent or intervening normal tissues. Linear structures (like the spinal cord) and tubular structures (like the bowels) are commonly called "serially functioning tissues" akin to series electrical circuits because their function is disrupted if there is a defect anywhere along their pathways.
Arm/Group | Image Guided Hypfractioned Radiation Treatment
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female participants | 16
  male participants | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Time Taken to Induce Primary Tumor Control
Description: The primary objective is to improve primary tumor local control of eligible LACC using SABR as the mechanism for delivering boost therapy to 85% at 2 years post treatment
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: daya
Groups:
- SABR Boost Therapy: SABR Boost Therapy
Arm/Group | SABR Boost Therapy
Number analyzed (Participants) | 16
daya | 55 [55 to 77]

ADVERSE EVENTS:
Time Frame: The AE's were collected up to 90 days
Groups:
- SABR Boost Therapy: SABR Boost Therapy: a. Initial Pelvic (+/- Para-aortic) fractionated external beam Radiation with 45 Gy to combined PTV with a boost to 55Gy for PET positive/CT enlarged nodes; b. Image Guided Hypofractionated Radiation Treatment boost to Cervix High risk CTV/PTV 28GY/4 fx.
  Patients will receive 4 fractions of 7 Gy each via stereotactic body radiation as boost therapy to a volume that encompasses the cervical tumor. A minimum of 40 hours should separate each treatment.
Arm/Group | SABR Boost Therapy
All-Cause Mortality (participants affected / at risk) | 7/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SABR Boost Therapy (N=16)
Death (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (16) — 1 patient developed grade 2 rectal bleeding. Of the grade 3 toxicities, 1 patient had grade 3 diarrhea consisting of greater than 8 stools over baseline per day which occurred 32 days after treatment and lasted two days.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SABR Boost Therapy (N=16)
Rectal Fistula (Gastrointestinal disorders) | 1
Rectal Bleeding (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Vaginal Bleeding (Reproductive system and breast disorders) | 1
Rectal Proctitis (Gastrointestinal disorders) | 1
Rectal Ulcer (Gastrointestinal disorders) | 1
Dysuria (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Vaginal Pain (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
Study was not completed .the total number of accrual was not met

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02045433/Prot_SAP_000.pdf